CLINICAL TRIAL: NCT04744545
Title: Randomized Controlled Trial of Adjunctive Curcumin and the Meru Health Program for Adults With Depression
Brief Title: RCT of Adjunctive Curcumin and the Meru Health Program
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Meru Health, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: #20-MERU-106
Record Dates: First submitted 2021-01-25; First posted 2021-02-09 (Actual); Last update posted 2023-07-13 (Actual); Status verified 2023-07

CONDITIONS: Depression
MeSH Terms: conditions — Depression | interventions — Curcumin

STUDY DESIGN:
Intervention Model Description: Randomized controlled trial with two study groups.
Who Masked: Outcomes Assessor
Masking Description: Outcomes assessors will not have information about each participant's study group.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Meru Health Program plus adjunctive curcumin (MHP-CUR) (Experimental): Meru Health Program (12 week program) with participants taking 2 turmeric supplements (1500mg/day) curcumin.
  Interventions: Behavioral: Meru Health Program; Dietary Supplement: Curcumin
- Meru Health Program (MHP-ONLY) (Active Comparator): Meru Health Program (12 week program)
  Interventions: Behavioral: Meru Health Program

INTERVENTIONS:
Behavioral: Meru Health Program — 12 week evidence-based mental health intervention overseen by a licensed clinical therapist delivered via Smartphone app
Dietary Supplement: Curcumin — 1500mg/day curcumin plus black pepper to aid absorption
  Arms: Meru Health Program plus adjunctive curcumin (MHP-CUR)

SUMMARY:
This is a randomized controlled trial (RCT) to compare the Meru Health Program plus adjunctive curcumin (MHP-CUR) versus Meru Health Program only (MHP-ONLY) for adults with depression. Meru Health is a 12-week integrative treatment program based on several evidence-based practices and overseen by licensed clinical therapists that is delivered via a Smartphone app. The primary objective of the study is to determine the feasibility, initial efficacy (depressive symptoms), and potential harms of taking adjunctive curcumin supplementation during the 12-week MHP among adults with depression. Secondary objectives include comparing changes in inflammation biomarkers, anxiety, worker productivity, and burnout that occur during the program between those in MHP-CUR and MHP-ONLY.

DETAILED DESCRIPTION:
This is a randomized controlled trial (RCT) to compare the Meru Health Program plus adjunctive curcumin (MHP-CUR) versus Meru Health Program only (MHP-ONLY) for adults with depression. Meru Health is a 12-week integrative treatment program based on several evidence-based practices and overseen by licensed clinical therapists that is delivered via a Smartphone app. The primary objective of the study is to determine the feasibility, initial efficacy (depressive symptoms), and potential harms of taking adjunctive curcumin supplementation during the 12-week MHP among adults with depression. Secondary objectives include comparing changes in inflammation biomarkers, anxiety, worker productivity, and burnout that occur during the program between those in MHP-CUR and MHP-ONLY.

This feasibility study will use a randomized controlled trial of up to 60 adult patients with depression. Patients will be recruited through Facebook ads, complete online and telephone/Zoom screening and, if eligible, invited to participate in the 12-week Meru Health program. One group will be randomized to being in the MHP plus receiving curcumin supplementation (MHP-CUR) and the other will be randomized to being in the MHP only (MHP-only). The MHP overseen by a licensed therapist who is available to the participant as needed via text messaging and, when requested, telephone. The program is delivered via an app downloaded to the user's Smartphone made available via email. The lab orders will be sent to each patient's Ultalabs center of choice or, if preferred, done in the patient's home. All study participants (in both groups) will be asked to get their blood drawn before starting the program, 6 weeks into the program, and just after the 12-week program. Two vials of blood will be taken at each visit, one to test for high sensitivity-CRP (hs-CRP) levels and the other to test for interleukin (IL-6) levels. 2ml of serum is needed for each vial. Patients in both groups will receive a wearable HRVB device via US mail; patients in the MHP-CUR group will also receive curcumin supplements via US mail. All non-laboratory study assessments will be made via the app and online via email.

ELIGIBILITY:
Inclusion Criteria:

* 18 years or older
* Patient presenting to the Meru Health online clinic
* Able to read and understand English
* Own a Smartphone
* Willing to commit to doing program practices for 10 minutes a day, 6 days a week for 12 weeks
* PHQ-9 of 10 or higher

Exclusion Criteria:

* Lifetime bipolar disorder or a psychotic disorder
* Possible cognitive impairment
* Substance use disorder in the past 3 months
* Active suicidal ideation with at least some intent to act
* Pregnant, breastfeeding, or desiring to become pregnant in the next 6 months
* Self-reported current suffering from a major medical illness including neurodegenerative/neuroinflammatory disorders, anemia, Alzheimer's disease, stroke, Parkinson's disease, or multiple sclerosis, autoimmune disorders, diabetes, inflammatory bowel disease, chronic obstructive pulmonary disease, asthma, coagulation disorder, cardiovascular disease, hypertension, chronic fatigue syndrome, fibromyalgia
* Self-reported current use of glucocorticoids, antibiotics, anticoagulant medications, antioxidant supplements (including curcumin), herbal supplements, or ω3 polyunsaturated fatty acids
* Self-reported past suffering from an infection or illness over the past month

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2021-02-01 (Actual); Primary Completion 2021-09-30 (Actual); Study Completion 2021-12-30 (Actual)

PRIMARY OUTCOMES:
Depression | 12 weeks
  Mean changes in the Patient Health Questionnaire, 9 item scale (PHQ-9) made during the program will be calculated. Scores range from 0 (no depression) to 27 (most severe depression)
Patient-reported adverse events | during the 12 week program
  The proportion of patients reporting at least one adverse event during the 12-week intervention will be reported.

SECONDARY OUTCOMES:
Anxiety | 12 weeks
  Mean changes in the Generalized Anxiety Disorder-7 item scale (GAD-7) will be reported. GAD-7 scores range from 0 (no anxiety) to 21 (most severe anxiety)
Burnout | 12 weeks
  The proportion of patients with changes in burnout will be reported. A validated, single-item burnout question will be used to assess burnout that has 5 response categoreis ranging from 1 (no burnout) to 5 (completed burned out) and dichotomized as <3 (no to low burnout) versus >=3 (at least moderate levels of burnout)
Worker productivity and activity impairment | 12 weeks
  The mean percent difference in each of the 4 subscales of the Worker Productivity and Activity Impairment (WPAI) scale will be reported. Subscales include absenteeism, presenteeism, overall worker productivity impairment, and impairment with daily activities and range from 0 (no impairment) to 100% (complete impairment).
Therapist rating | 12 weeks
  The proportion of patients who reported being satisfied with their program therapist will be reported as dichotmized by a 5-category scale that ranges from 1 (not at all satisfied) to 5 (extremely satisfied). Responses "1" and "2" (not at all satisfied and not satisfied) will be combined into a "not satisfied" dichotomous category and responses 2 (satisfied), 3 (very satisfied) and 4 (extremely satisfied) will be combined into a "satisfied" dichotomous category, with the proportion of patients falling into each category being reported.
Interleukin-6 | 12 weeks
  Mean changes in Interleukin-6 (IL-6) will be calculated for each participant to measure changes in inflammation made during the program.
High Sensitivity C Reactive Protein | 12 weeks
  Mean changes in high-sensitivity c reactive protein (hs-crp) will be calculated for each participant to measure changes in inflammation made during the program.

CONTACTS AND LOCATIONS:
Locations (1):
- Online, Denver, Colorado, United States

IPD SHARING:
Plan to Share IPD: Undecided